CLINICAL TRIAL: NCT04093531
Title: Pilot Trial of Ustekinumab for Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Ummara Shah, Assistant Professor of Medicine, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ustekinumab for PSS
Record Dates: First submitted 2019-08-05; First posted 2019-09-18 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Primary Sjögren Syndrome
Keywords: primary sjogren syndrome; PSS; SjS; Sjogren; Ustekinumab; SS
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Intervention Model Description: Up to 15 subjects will receive an infusion loading dose of 6 mg/kg of ustekinumab at baseline, and 90 mg of ustekinumab subcutaneously at week 4, week 12 and week 20. Subjects will be followed for 24 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ustekinumab (Experimental): All subjects will receive an intravenous loading dose of 6 mg/kg at their baseline visit. 650mg acetaminophen and 60mg allegra will be given as premedication to the infusion. All patients will receive 90mg ustekinumab by a subcutaneous injection at all subsequent dosing visits. Subcutaneous injections do not require any premedication. Drug will be administered by qualified personnel.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Up to 15 subjects will receive an infusion loading dose of 6 mg/kg of ustekinumab at baseline, and 90 mg of ustekinumab subcutaneously at week 4, week 12 and week 20. Subjects will be followed for 24 weeks.

SUMMARY:
This pilot study will make a preliminary determination of the safety of ustekinumab in patients with Primary Sjogren's Syndrome (PSS) and assess the response of systemic measures of inflammation (biomarkers).

DETAILED DESCRIPTION:
This is a single-center, open label, pilot trial of ustekinumab in patients with Primary Sjögren's Syndrome (PSS). Up to 15 subjects will receive an infusion loading dose of 6 mg/kg of ustekinumab at baseline, and 90 mg of ustekinumab subcutaneously at week 4, week 12 and week 20. Subjects will be followed for 24 weeks.

ELIGIBILITY:
A subject who has met all of the following criteria is eligible for participation in the study:

* Has provided written informed consent
* Between the ages of 18-75 years (inclusive)
* Body weight ≥ 40 kg
* Meets the 2016 ACR EULAR criteria (score >4)

  * 3 points- Labial salivary gland with focal lymphocytic sialadenitis and focus score of >1 foci/4 mm2‡
  * 3 Points- Anti-SSA/Ro positive
  * 1 Point- Ocular Staining Score >5 in at least 1 eye
  * 1 Point- Schirmer's test <5 mm/5 minutes in at least 1 eye
  * 1 Point- Unstimulated whole saliva flow rate <0.1 ml/minute
* If taking prednisone (or equivalent corticosteroid), the dose must be ≤ 10 mg/day and stable for at least 4 weeks prior to baseline visit
* If taking hydroxychloroquine, the dose must be stable for at least 12 weeks prior to baseline.
* If taking a cholinergic stimulant (e.g. pilocarpine, cevimeline), the dose must be stable for at least 4 weeks prior to baseline.
* If a male of reproductive potential, must agree to practice two highly effective forms of contraception during the study (one of which must be a barrier method) and be able to continue contraception for 20 weeks after his last dose of study agent Subject must also agree not to donate sperm up to 20 weeks after his last dose of study agent.
* If a female of childbearing potential, must agree to practice two highly effective forms of contraception during the study (one of which must be a barrier method) and able to continue contraception for 20 weeks after her last dose of study agent.

A subject who meets any of the following criteria is disqualified from participation in the study:

* Has a chronic or persistent infection that might be worsened by immunosuppressive treatment (e.g., HIV, hepatitis B, hepatitis C, or tuberculosis).
* History of untreated TB or positive QuantiFERON TB-Gold during screening period. If a subject has previously received an adequate course of therapy for either latent (9 months of isoniazid in a locale where rates of primary multi-drug resistant TB infection are <5%) or active TB infection, a QuantiFERON TB-Gold test need not be obtained, but a chest radiograph or other appropriate image must still be obtained if not done so within the prior 3 months.
* History of recurrent significant infections or occurrence of a serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within twelve weeks prior to Day 0.
* Active symptomatic infection within two weeks prior to Day 0.
* Receipt of live vaccine within four weeks prior to Day 0.
* History or presence of primary or secondary immunodeficiency.
* History of any life-threatening allergic reactions to pilocarpine or any components of ustekinumab. Pilocarpine will be used to stimulate salivary flow in order to assess flow rate.
* Is currently pregnant or nursing.
* Concurrent use of anticholinergic agents, such as tricyclic antidepressants, antihistamines, phenothiazines, antiparkinsonian drugs, anti-asthmatic medications, or gastrointestinal (GI) medications that cause xerostomia in more than 10% of patients.
* Treatment with any of the following within the defined period prior to the screening and Day 0 visits:

  * 12 months for rituximab
  * 24 weeks for cyclophosphamide
  * 8 weeks for azathioprine, cyclosporine, methotrexate, and mycophenolate mofetil
  * 4 weeks for intravenous immunoglobulin
  * 4 weeks for etanercept
  * 8 weeks for adalimumab
  * 12 weeks for infliximab
  * 8 weeks Golimumab
  * 8weeks Certolizumab pegol
  * 16 weeks Abatacept
  * 4 weeks Tocilizumab SQ
  * 16 weeks Tocilizumab IV
  * 4 weeks Tofacitinib and Tofacitinib XR
* Prednisone (or equivalent corticosteroid) > 10 mg/day.
* A definite diagnosis of RA, SLE, systemic sclerosis, or dermatomyositis.
* A history of alcohol or substance abuse.
* A history of head and neck radiation therapy, sarcoidosis, or graft-versus-host disease.
* A history of malignancy, except for a resected basal or major squamous cell carcinoma, cervical dysplasia, or in situ cervical cancer Grade I, within the last five years.
* Abnormal laboratory results for the following parameters at the baseline visit:

  * Absolute neutrophil count (ANC): < 1500/mm3
  * Platelets: < 100,000/mm3
  * Hemoglobin: < 9 grams (g)/deciliter (dL)
  * Serum creatinine: ≥ 2.0 mg/dL
  * AST: > 1.5x upper limit of normal
  * ALT: > 1.5x upper limit of normal.
* A psychiatric disorder rendering the subject incapable of providing informed consent.
* Plans for foreign travel to countries other than Canada or Western Europe within the treatment period.
* Inability or unwillingness to follow the protocol
* Any condition or treatment that, in the opinion of the investigator, places the subject at an unacceptable risk as a participant in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ummara Shah, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 subjects were consented. 4 failed screening.
Period: Overall Study
Arm/Group | Ustekinumab
Started | 12
Completed | 8
Not Completed | 4
Not completed — failed screening | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ustekinumab
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 47.3 [27 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in The European League Against Rheumatism (EULAR) Sjogren's Syndrome Patient Reported Index (ESSPRI) Score From Baseline to Week 24
Description: The primary endpoint is a well-established, patient reported questionnaire for use in PSS, the ESSPRI. The ESSPRI is composed of 3 scales - dryness, fatigue, and pain. Each scale is measured 0 - 10, 0 being no symptoms, 10 being maximal imaginable dryness, fatigue or pain. The total score is the mean score of the three scales which ranges from 0- 10. Baseline ESSPRI total score will be compared to week 24, end of treatment, ESSPRI total score.
Time Frame: baseline to 24 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ustekinumab
Number analyzed (Participants) | 8
score on a scale | -0.125 [-1 to 2]

2. Secondary Outcome: Change in the Short Form Health Survey (SF-36) Patient Reported Outcome Measure Between Day 0 and Week 24
Description: The SF-36 is a measure of health-related quality-of-life. It's a 36-item patient-reported questionnaire that covers 8 health domains. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state. Changes in total scores in each domain from BL to week 24 will be measured for physical function, energy/fatigue, pain and general health.
Time Frame: baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ustekinumab
Number analyzed (Participants) | 8
score on a scale
  physical function | 11.1 (8.9)
  energy/fatigue | 7.5 (17.9)
  pain | 5.25 (15.5)
  general health | 0.6 (20.1)

3. Secondary Outcome: Change in Mean Serum Biomarkers of Inflammation From Baseline to Week 24
Description: To determine whether the standard dosing schedule for ustekinumab lowers serum biomarkers of inflammation in patients with PSS blood will be collected at baseline and week 24 for the following mechanistic studies: Serum levels of TNFα, IL-6, IL17, IL17A, IL17F, IL22, IL12, IL23, BAFF, B and T cell, blood interferon signature.
Time Frame: baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ustekinumab
Number analyzed (Participants) | 8
pg/mL
  IFNa2 | 6.984 (0.2922)
  IL12p40 | 12.62 (0.0893)
  IP-10 | 111.3 (0.6145)
  IL-17F | 0.02175 (0.3683)
  IFNg | -0.3912 (0.9705)
  IL12p70 | 3.054 (0.0204)
  IL-13 | 1.689 (0.6965)
  IL17A | -1.236 (0.4774)
  IL-22 | 0.2963 (0.2742)
  IL-23 | 1.456 (0.1801)
  IL-6 | 2.411 (0.2198)
  TNFa | 1.374 (0.1252)

4. Secondary Outcome: Total Score of the EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI)
Description: The ESSDAI is a disease activity measurement that has 12 domains. The score of each domain is the product of the weight of the domain by the level of activity. Lower numbers indicate less activity. The total score is the sum of the score of all domains. The total score ranges from 0-123. Mean scores at baseline and week 24 are reported.
Time Frame: 24 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ustekinumab
Number analyzed (Participants) | 8
score on a scale
  Baseline | 2.86 (3.563)
  Week 24 | 1.75 (1.5811)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Ustekinumab
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab (N=8)
bilateral leg pain (Musculoskeletal and connective tissue disorders) | 1
chest heaviness (General disorders) | 1
Conjunctival Hemorrhage in right eye (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Double Vision (Eye disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Enlarged lymph node (Blood and lymphatic system disorders) | 2
Erythema right eyebrow (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 2
headache (Nervous system disorders) | 1
abdominal pain (Gastrointestinal disorders) | 1
menopause (Reproductive system and breast disorders) | 1
muscle tenderness right shoudler (Musculoskeletal and connective tissue disorders) | 1
nausea (Gastrointestinal disorders) | 5
right ankle sprain (Injury, poisoning and procedural complications) | 1
scalp rash (Skin and subcutaneous tissue disorders) | 1
sinus infection (Infections and infestations) | 1
vertigo (Ear and labyrinth disorders) | 1
worsening GI reflux (Gastrointestinal disorders) | 1
worsening hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was under enrolled and therefore not powered to show an effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT04093531/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT04093531/ICF_001.pdf